CLINICAL TRIAL: NCT04750135
Title: Assessment of Metformin as Adjuvant Therapy in Patients With Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Doaa abdelaziz, Lecturer at pharmacy practice department, FUE, Egypt, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-2019
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): participants will receive placebo for 8 consecutive weeks in addition to the standard therapy
  Interventions: Drug: Placebo
- Metformin group (Experimental): participants will receive 500 mg Metformin TID for 8 consecutive weeks in addition to the standard therapy
  Interventions: Drug: metformin 500 mg TID Oral Tablet

INTERVENTIONS:
Drug: metformin 500 mg TID Oral Tablet — biguanides derivatives
  Other Names: Glucophage XR
  Arms: Metformin group
Drug: Placebo — Placebo
  Arms: Control group

SUMMARY:
Brief Summary:

This is a randomized, controlled study evaluating metformin tablets administered daily for 8 weeks. The purpose of the study is to evaluate the efficacy and safety of metformin in the treatment of mild to moderately active ulcerative colitis. Disease activity will be measured using Mayo score for ulcerative colitis activity. Calculation of the score requires patients to undergo colonoscopy at the start of the study and at week 8.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild or moderate ulcerative colitis newly diagnosed by colonoscopy and biopsy according to Mayo endoscopic scoring of ulcerative colitis.
2. Adults (males and/or females) with age range from 18 to 65 years old.
3. Patients on treatment with 5-aminosalisylic acid (5-ASA)

Exclusion Criteria:

1. Patients with severe ulcerative colitis according to Mayo endoscopic scoring of ulcerative colitis.
2. Treatment with systemic or rectal steroids.
3. Treatment with immunosuppressants.
4. Previously failed treatment with a sulphasalazine.
5. Known hypersensitivity to any of study drugs.
6. Hepatic and renal dysfunction.
7. Pregnancy and lactation.
8. History of colorectal carcinoma.
9. History of complete or partial colectomy.
10. Current or previous treatment with metformin for females with polycystic ovarian syndrome.
11. Patients with diabetes mellitus
12. Patients with history of lactic acidosis
13. Patients with disease states associated with hypoxemia including cardiorespiratory insufficiency
14. Positive stool culture for enteric pathogens, positive stool ova and parasite exam.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-07 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference between the two groups in the expression of colonic (NF)-κB proteins. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, PhD, Principal Investigator — Mansoura University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hegazy SK, El-Bedewy MM. Effect of probiotics on pro-inflammatory cytokines and NF-kappaB activation in ulcerative colitis. World J Gastroenterol. 2010 Sep 7;16(33):4145-51. doi: 10.3748/wjg.v16.i33.4145. PMID 20806430
- [Background] Lewis JD, Lichtenstein GR, Deren JJ, Sands BE, Hanauer SB, Katz JA, Lashner B, Present DH, Chuai S, Ellenberg JH, Nessel L, Wu GD; Rosiglitazone for Ulcerative Colitis Study Group. Rosiglitazone for active ulcerative colitis: a randomized placebo-controlled trial. Gastroenterology. 2008 Mar;134(3):688-95. doi: 10.1053/j.gastro.2007.12.012. Epub 2007 Dec 7. PMID 18325386
- [Background] Samman FS, Elaidy SM, Essawy SS, Hassan MS. New insights on the modulatory roles of metformin or alpha-lipoic acid versus their combination in dextran sulfate sodium-induced chronic colitis in rats. Pharmacol Rep. 2018 Jun;70(3):488-496. doi: 10.1016/j.pharep.2017.11.015. Epub 2017 Nov 24. PMID 29653414